CLINICAL TRIAL: NCT02733250
Title: A Phase I/II Study of Pembrolizumab in Combination With Nab-Paclitaxel in Patients With Unresectable Stage III or Stage IV Non-Small Cell Lung Carcinoma
Brief Title: Pembrolizumab With Nab-Paclitaxel in Non-Small Cell Lung Cancer
Acronym: URCOH-PMS-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Merck Canada Inc. (Industry); Celgene (Industry); Jewish General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE15.274
Record Dates: First submitted 2016-03-15; First posted 2016-04-11 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
Keywords: NSCLC; Pembrolizumab; Nab-paclitaxel
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Nab-Paclitaxel (Other): Phase I will determine the recommended Phase II dose (RP2D) of nab-paclitaxel when given in combination with pembrolizumab. Escalation for nab-paclitaxel will be conducted following a "3+3" design. First cohort of 3 patients will receive nab-paclitaxel on Days 1 and 8 at a dose of 100 mg/m2 intravenous (IV) in combination with pembrolizumab at 200 mg IV every 3 weeks. If no dose limiting toxicities (DLT) occur, the dose of nab-paclitaxel will be escalated to 100 mg/m2 on Days 1, 8 and 15 every 3 weeks. The dose of pembrolizumab will remain the same. If no DLTs occur, dose level 2 will be defined as the RP2D. In the Phase II, pembrolizumab will be administered at 200 mg IV every 3 weeks and nab-paclitaxel will be administered at the RP2D.
  Interventions: Biological: Pembrolizumab; Drug: Nab-Paclitaxel

INTERVENTIONS:
Biological: Pembrolizumab — 200mg IV Day 1 of each 21 cycles
  Other Names: Keytruda
Drug: Nab-Paclitaxel — 100mg/m2 IV Day 1, 8 and 15 of every 21 day cycles
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to determine the optimal dose of nab-paclitaxel to be safely administered in combination with pembrolizumab in patients with advanced inoperable non-small cell lung cancer. The study is also aimed at evaluating the efficacy of the combination therapy.

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, proof of concept study of nab-paclitaxel administered in combination with pembrolizumab in patients with advanced non-small cell lung cancer (NSCLC).

Part 1 of the study will assess the dose limiting toxicity (DLT) of nab-paclitaxel in combination with a fixed dose of pembrolizumab (200 mg administered on day 1 of each 21 day cycle). Dose escalation for nab-paclitaxel will be conducted according to the "3+3 design" until the recommended phase 2 dose (RP2D) is determined.

Part 2 of the study will evaluate the administration of pembrolizumab at a dose of 200 mg every 3 weeks in combination with nab-paclitaxel at the RP2D. Determining the RP2D will classify the treatment combination as safe and allow for an expansion of the study population, which will ultimately lead to further assessments of safety and tolerability as well as an evaluation of the anti-tumoral effect of the proposed treatment combination.

Using Simon's optimal 2-stage design for Phase II clinical trials, we determined that a sample size of 36 patients would be adequate to test the proposed hypothesis.

The primary efficacy analysis of overall response rate (ORR) will be interpreted as follows: 1) if less than 9 partial response (PR) or complete response (CR) are recorded, the combination of nab-paclitaxel and pembrolizumab provides less than additive effects and is not likely to be clinically superior compared to pembrolizumab alone based on an ORR assessment; 2) however, if 9 or more PR or CR are recorded, the treatment combination warrants further clinical study. This could take the form of an extended phase II (to reach the 97 patients calculated from the model) or a phase III study.

Treatment will continue until disease progression (as per RECIST 1.1), unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, investigator's noncompliance with trial treatment or procedures requirements, the subject receives 24 months of uninterrupted treatment or 35 administrations of study medication (whichever is later), or administrative reasons.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have unresectable stage III (not eligible to curative-intent chemo-radiotherapy) or stage IV non-small cell lung cancer (NSCLC) according to the Clarification of Malignant Tumours (TNM) staging system for lung cancer (7th edition).
* Patients must be willing to undergo a biopsy procedure before the start of treatment unless these two conditions are met: 1) the biopsy must have been conducted after progression or intolerance to systemic first-line treatment as stated in criteria 7 and; 2) all the planned correlative analyses can be conducted on the available tissue.
* Have measurable/evaluable disease based on the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Have an Eastern Cooperative Oncology Group (ECOG) of 0 or 1.

Exclusion Criteria:

* Has a known epidermal growth factor receptor (EGFR) sensitizing (activating) mutation and/or anaplastic lymphoma kinase (ALK) translocation.
* Has an unknown EGFR and ALK status.
* Has received prior therapy with paclitaxel or docetaxel for NSCLC.
* Has received systemic steroid therapy within three days prior to the first dose of study treatment or receiving any other form of systemic immunosuppressive medication.
* Has a history of allogeneic tissue/solid organ transplant.
* Has prior systemic cytotoxic chemotherapy, antineoplastic biological therapy, major surgery within 3 weeks of the first dose of study drug; received prior tyrosine kinase inhibitor therapy or completed palliative radiotherapy within 7 days of the first dose of study drug.
* Has an active infection requiring systemic therapy.
* Has received prior therapy with an anti-programmed cell death protein 1 (PD-1), including pembrolizumab, anti-programmed cell death protein ligand 1 (anti-PD-L1), anti-programmed cell death protein ligand 2 (anti-PD-L2), anti-tumor necrosis factor (CD137), or anticytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug targeting immune checkpoint pathways).
* Has had any other malignancy within 5 years prior to the start of therapy. Exceptions are malignancies with a negligible risk of metastasis or death (e.g., expected 5-year overall survival (OS) > 90%).
* Has known active central nervous system (CNS) metastases or leptomeningeal involvement.
* Has active autoimmune disease (or documented history), or a syndrome that requires systemic corticosteroids or immunosuppressive agents (patients with auto-immune thyroid disease, vitiligo or well controlled type 1 diabetes mellitus are eligible).
* Has known history or active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Women of childbearing potential who is unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of nab-paclitaxel in combination with pembrolizumab as measured by incidence of drug related adverse events (AEs), serious drug related AEs, dose-limiting toxicities. | Safety follow-up will be maintained up to 90 days following the administration of the last study-drug dose.
  Safety analysis will be based on subjects who experienced toxicities as defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who received at least one dose of pembrolizumab and nab-paclitaxel, including serious adverse events (SAEs) and event of clinical interest (ECIs).
Objective Response Rate (ORR) | up to 56 months
  Defined as the proportion of patients with best overall response or either complete response or partial response, which will be recorded based on the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or the Immune related response criteria (irRC).

CONTACTS AND LOCATIONS:
Overall Officials: Normand Blais, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Canada (2):
  - Centre hospitalier de l'université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591